CLINICAL TRIAL: NCT01151150
Title: The Phenomenon of "Chronic Lyme"; an Observational Study
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Unn Ljøstad PhD, MD, Sorlandet Hospital HF
Other Study IDs: Chronic Lyme
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Lyme Borreliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, CSF
Oversight: Data Monitoring Committee: No

SUMMARY:
The current study is set up to chart clinically and laboratory findings in Norwegian patients with symptoms attributed by themselves or their doctor to ongoing chronic Bb infection. Objectives is to assess laboratory findings in relation to established diagnostic criteria and to form a picture of the burden of symptoms and illness perception in this group of patients. The study is essentially exploratory, and is supposed to raise rather than to test hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms attributed by themselves or their doctor to ongoing chronic Bb infection

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible if they themselves or their physician suspected that they suffer from ongoing chronic Bb infection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sølandet Hospital HF, Kristiansand, Norway